CLINICAL TRIAL: NCT02099201
Title: A Single-center, Double-blind, Parallel-group, Randomized, Placebo-controlled, Multiple-ascending Oral Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ACT-389949 in Healthy Subjects
Brief Title: Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ACT-389949 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: AC-073-102
Record Dates: First submitted 2014-03-26; First posted 2014-03-28 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Healthy Subjects
Keywords: ACT-389949
MeSH Terms: interventions — ACT-389949

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Group A1 (Experimental): Ten subjects will receive ACT-389949 40 mg and 3 subjects will receive placebo, once a day for 9 days Medication will be administered orally, in the morning, following an overnight fast.
  Interventions: Drug: ACT-389949 40 mg; Drug: Placebo
- Group A2 (Experimental): Ten subjects will receive ACT-389949 (Predicted to be 200 mg) and 3 subjects will receive placebo, once a day for 9 days Medication will be administered orally, in the morning, following an overnight fast.
  Interventions: Drug: ACT-389949 200 mg; Drug: Placebo
- Group A3 (Experimental): Ten subjects will receive ACT-389949 (Predicted to be 800 mg) and 3 subjects will receive placebo, once a day for 9 days Medication will be administered orally, in the morning, following an overnight fast.
  Interventions: Drug: ACT-389949 800 mg; Drug: Placebo
- Group B1 (Experimental): Ten subjects will receive ACT-389949 200 mg and 3 subjects will receive placebo, every 3 days for 13 days (a total of 5 doses), administered orally, in the morning, following an overnight fast.
  Interventions: Drug: ACT-389949 200 mg; Drug: Placebo
- Group B2 (Experimental): Ten subjects will receive ACT-389949 (provisionally 200 mg) and 3 subjects will receive placebo, every 2 days for 9 days (a total of 5 doses), administered orally, in the morning following an overnight fast. The actual dose will depend on the emerging data from Group B1.
  Interventions: Drug: ACT-389949 200 mg; Drug: Placebo
- Group C1 (Experimental): 10 subjects will receive ACT-389949 and 3 subjects on placebo. The actual dose will depend on the emerging data from the previous groups but will be within the dose range or lower than the dose range tested in Part A. The dosing schedule will be one of those already tested in Part A and/or Part B.
  Interventions: Drug: ACT-389949 (Group C1 dose to be selected); Drug: Placebo
- Group C2 (Experimental): 10 subjects will receive ACT-389949 and 3 subjects on placebo. The actual dose will depend on the emerging data from the previous groups but will be within the dose range or lower than the dose range tested in Part A. The dosing schedule will be one of those already tested in Part A and/or Part B.
  Interventions: Drug: ACT-389949 (Group C2 dose to be selected); Drug: Placebo

INTERVENTIONS:
Drug: ACT-389949 40 mg
  Arms: Group A1
Drug: ACT-389949 200 mg — Predicted dose
  Arms: Group A2; Group B1; Group B2
Drug: ACT-389949 800 mg — Predicted dose
  Arms: Group A3
Drug: ACT-389949 (Group C1 dose to be selected)
  Arms: Group C1
Drug: ACT-389949 (Group C2 dose to be selected)
  Arms: Group C2
Drug: Placebo

SUMMARY:
This is a single-center, double-blind, parallel-group, randomized, placebo-controlled, multiple-ascending oral dose study to investigate the safety, tolerability, pharmacokinetics, and pharmacodynamics of ACT-389949 in healthy subjects.

Part A of the study will evaluate the safety and tolerability following once a day oral dosing of ACT-389949 for 9 days and investigate ACT-389949 pharmacokinetics and pharmacodynamics.

Part B of the study will evaluate the safety and tolerability of ACT-389949 following a maximum of two different oral dosing regimens: ACT-389949 given either every 3 days for 13 days or every 2 days for 9 days (5 doses for each regimen).

Part C of the study, if required, will provide additional information to that obtained from Parts A and B in terms of safety, tolerability, pharmacokinetics, and pharmacodynamics of ACT-389949.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in local language.
* Healthy Caucasian male subjects and female subjects of non-childbearing potential.
* Men with female partners of childbearing potential must agree to use 2 reliable methods of contraception from first drug administration up to a minimum of 90 days after the end of treatment.
* Male subjects must agree not to donate sperm from the first drug administration until 90 days after the end of treatment.
* Non-smokers, defined as never smoked or achieved cessation ≥ 12 months prior to screening.
* Body mass index of 18.0 to 28.0 kg/m^2 (inclusive) at screening.
* No clinically significant findings on the physical examination at screening.
* Negative results from urine alcohol and drug screen at screening and on Day -1.
* Systolic blood pressure 100-145 mmHg, diastolic blood pressure 50-90 mmHg, and pulse rate 45-90 beats per minute (inclusive) measured at screening.
* 12-Lead electrocardiogram without clinically relevant abnormalities at screening.
* Body temperature 35.5-37.7 °C at screening and prior to first dosing.
* C-reactive protein (CRP) and total and differential white blood cell (WBC)count within the local laboratory normal ranges at screening and on Day -1.
* Hematology, coagulation, clinical chemistry, and urinalysis results (other than total differential WBC and CRP), not deviating to a clinically relevant extent from the normal local laboratory range(s) at screening.
* Forced expiratory volume in 1 second (FEV1) ≥ 80% of predicted, FEV1 / Forced vital capacity ≥ 70%.
* Subjects must be able to provide adequate sputum following induction with hypertonic saline at screening.
* Able to communicate well with the investigator, in the local language, and to understand and comply with the requirements of the study.
* Able to stay in the unit for the entire duration required and undertake all study related procedures.

Exclusion Criteria:

* Circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.
* History or clinical evidence of any disease and/or existence of any surgical or medical condition which might interfere with the absorption, distribution, metabolism or excretion of the study drug.
* Previous history of fainting, collapse, syncope, orthostatic hypotension, or vasovagal reactions.
* Veins unsuitable for intravenous puncture on either arm.
* Loss of 250 mL or more of blood or blood donation, within 3 months prior to screening.
* Known allergic reactions or hypersensitivity to any excipient of the drug formulation(s).
* Previous exposure to ACT-389949.
* Exposure to lipopolysaccharide within the last year.
* Treatment with another investigational drug within 3 months prior to screening or participation in more than 4 investigational drug studies within 1 year prior to screening.
* History or clinical evidence of alcoholism or drug abuse within the 3-year period prior to screening.
* Excessive caffeine consumption.
* Use of regular medication or therapy (including vaccines) or over-the-counter medications within 2 weeks prior to first study drug administration or 5 half-lives of the medication, whichever is longer.
* Positive results from the hepatitis serology, except for vaccinated subjects or subjects with past but resolved hepatitis, at screening.
* Positive results from the human immunodeficiency virus serology at screening.
* Vaccinations within the previous 6 months or foreign travel to areas within the last 6 months where infectious diseases are prevalent.
* Signs or symptoms suggestive of infection within 2 weeks prior to study screening and between screening and dosing.
* Signs of respiratory tract infections within 2 weeks prior to screening and between screening and dosing.
* History of atopic allergy.
* Hay fever, if within active season.
* Chronic diseases including those with recurring periods of flare-ups and remission.
* Legal incapacity or limited legal capacity at screening.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2012-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline up to end of study in supine systolic blood pressure | Up to 13 days
  Blood pressure will be measured using an automatic oscillometric device, always on the dominant arm (i.e., dominant arm right = writing with right hand)
Change from baseline up to end of study in supine diastolic blood pressure | Up to 13 days
  Blood pressure will be measured using an automatic oscillometric device, always on the dominant arm (i.e., dominant arm right = writing with right hand)
Change from baseline up to end of study in pulse rate | Up to 13 days
  Pulse rate will be measured using an automatic oscillometric device, always on the dominant arm (i.e., dominant arm right = writing with right hand)
Change from baseline up to end of study in body temperature | Up to 13 days
  Body temperature will be measured in the ear, where possible using the same thermometer(s) for all the subjects throughout the study.
Change from baseline up to end of study in body weight | Up to 13 days
  Body weight will be measured where possible using the same weighing scale for all subjects throughout the study. The weighing scale should have a precision of at least 0.5 kg.
Change from baseline up to end of study in PQ/PR interval (time interval from the beginning of the P wave to the beginning of the QRS complex) | Up to 13 days
  PQ/PR interval will be determined from standard 12-lead electrocardiogram (ECG) recorded in the supine position, after a 5-minute period of resting.
Change from baseline up to end of study in QRS duration (time interval from the beginning of the Q wave to the end of the S wave) | Up to 13 days
  QRS duration will be determined from standard 12-lead ECG recorded in the supine position, after a 5-minute period of resting.
Change from baseline up to end of study in QT interval (time interval from beginning of the Q wave until end of the T wave) | Up to 13 days
  QT interval will be determined from standard 12-lead ECG recorded in the supine position, after a 5-minute period of resting.
Change from baseline up to end of study in QTcB interval according to Bazett's correction (QTcB) | Up to 13 days
  QTcB interval will be determined from standard 12-lead ECG recorded in the supine position, after a 5-minute period of resting. The QTcB interval is the QT interval corrected for heart rate with Bazett's formula (QTcB = QT/RR^0.5 where RR is 60/heart rate)
Change from baseline up to end of study in QTcF interval according to Fridericia's correction (QTcF) | Up to 13 days
  QTcF interval will be determined from standard 12-lead ECG recorded in the supine position, after a 5-minute period of resting. The QTcB interval is the QT interval corrected for heart rate with Fridericia's formula (QTcB = QT/RR^0.33 where RR is 60/heart rate)
Frequency of treatment-emergent ECG abnormalities from baseline up to end of study | Up to 13 days
  Treatment-emergent abnormalities will be determined from standard 12-lead ECGs recorded in the supine position, after a 5-minute period of resting.

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve of ACT-389949 during the dosing interval (AUCτ,Dayx) | Up to 13 days
  Blood samples for pharmacokinetic analysis will be taken immediately prior to dosing with ACT-389949, and at various time points after dosing. AUCτ,Dayx will be calculated according to the linear trapezoidal rule using the measured concentration-time values above the lower limit of quantification during the dosing interval.
Maximum plasma ACT-389949 concentration during the dosing interval (Cmax,Dayx) | Up to 13 days
  Blood samples for pharmacokinetic analysis will be taken immediately prior to dosing with ACT-389949, and at various time points after dosing. Cmax,Dayx will be calculated on the basis of the blood sampling time points.
Average plasma ACT-389949 concentration during the dosing interval (Cav,Dayx) | Up to 13 days
  Blood samples for pharmacokinetic analysis will be taken immediately prior to dosing with ACT-389949, and at various time points after dosing. Cav,Dayx will be calculated by dividing AUCτ,Dayx by the dosing interval.
Time to reach maximum plasma ACT-389949 concentration (tmax,Dayx) | Up to 13 days
  Blood samples for pharmacokinetic analysis will be taken immediately prior to dosing with ACT-389949, and at various time points after dosing. tmax,Dayx will be calculated on the basis of the blood sampling time points.
Accumulation index (AI) of ACT-389949 | Up to 13 days
  Blood samples for pharmacokinetic analysis will be taken immediately prior to dosing with ACT-389949, and at various time points after dosing. The AI will be calculated as follows: AUCτDayx / AUCτDay1.
Trough concentration (Ctrough,Dayx) of ACT-389949 | Up to 13 days
  Blood samples for pharmacokinetic analysis will be taken immediately prior to dosing with ACT-389949, and at various time points after dosing. Ctrough,Dayx of ACT-389949 will be taken directly from the measured plasma concentration-time values.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Mackie, MSc, Study Director — Actelion
Locations (1):
- Celerion, Belfast, United Kingdom